CLINICAL TRIAL: NCT03199443
Title: Pelvic Floor Electromyography Monitoring as Tool to Improve Patient Selection and Outcome - Standardization of Lead Placement for Sacral Neuromodulation.
Brief Title: Standardization of Lead Placement for Sacral Neuromodulation Part 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Donald Vaganée, Principal Investigator, Universiteit Antwerpen
Other Study IDs: B300201523497 Part 2
Record Dates: First submitted 2017-05-10; First posted 2017-06-27 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Overactive Bladder; Non Obstructive Urinary Retention
Keywords: Sacral neuromodulation; Electromyography; Pelvic floor
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Overactive bladder patients
  Interventions: Diagnostic Test: EMG pelvic floor
- Non Obstructive Urinary Retention patients
  Interventions: Diagnostic Test: EMG pelvic floor

INTERVENTIONS:
Diagnostic Test: EMG pelvic floor — EMG activity during tined lead test procedures will be monitored and the response on needle stimulation will be evaluated

SUMMARY:
Prospective observational study.

A substantial number of patients do not respond favourably to sacral neurostimulation (SNS) although clinically, they appear to have the same lower urinary tract (LUT) dysfunction characteristics as the good responders. This may be due to methodological issues (lead position) or patient selection. The purpose of this study is to improve and standardize lead position, in order to increase the patient response to test stimulation and to SNS treatment, and to decrease adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years and competent to provide consent
2. Minimum 3 months of self-reported OAB symptoms or self-reported obstructive lower urinary tract symptoms (LUTS) in addition to confirmed non-obstructive urinary retention on urodynamics.
3. Failed, or are not a candidate for more conservative treatment (i.e., pelvic floor training, biofeedback, behavioral modification, oral pharmacotherapy)
4. Willing to discontinue OAB medications for 2 weeks prior to the implant and for the entire study period
5. Able to thoroughly fill in all questionnaires, voiding diaries and office visits for device programming and clinical evaluations before the TLP, 3 weeks after TLP and 6 weeks, 6 months and 1 year after implantation of definitive IPG.

Exclusion Criteria:

1. Current of prior evidence of primary stress incontinence or mixed incontinence where the stress component overrides the urgency component
2. Any neurological condition that may interfere with normal bladder function, including stroke, multiple sclerosis, Parkinson's disease, clinically significant peripheral neuropathy, or spinal cord injury (e.g., paraplegia)
3. Urinary tract mechanical obstruction including but not limited to Benign Prostatic Hyperplasia (BPH)
4. Treatment of bladder or pelvic floor dysfunction with botulinum toxin (Botox ®) or surgery in past 12 months
5. Unable to toilet self and have and maintain good personal hygiene
6. Unable to provide clear, thoughtful responses to questions and questionnaires
7. Urinary tract, bladder or vaginal infection or inflammation
8. Hematuria, and absence of an elaborate diagnostic work-up
9. Severe or uncontrolled diabetes (A1C > 8, documented in the last 3 months) or diabetes with peripheral nerve involvement
10. Allergy to local anesthetic or adhesives
11. Bleeding disorder or on an anticoagulant that cannot be stopped for 3 days before the implant
12. Pregnant, lactating, planning to become pregnant, given birth in the past 12 months, or female of child-bearing potential and not practicing a medically-approved method of birth control
13. Skin lesions or compromised skin at the implant or stimulation site
14. Use of investigational drug or device therapy or participation in any study involving or impacting gynecologic, urinary or renal function within past 4 weeks
15. Passive implants (e.g., prostheses) are allowed, but no implanted metal should be at the Neurostimulator implant site
16. Knowledge of planned magnetic resonance imaging (MRI), diathermy, or high output ultrasonic exposure
17. Presence of a documented condition or abnormality that could compromise the safety of the patient
18. Any psychiatric or personality disorder at the discretion of the study physician
19. Interstitial cystitis or bladder pain syndrome as defined by the guidelines of the European Association of Urology (EAU).
20. Life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OAB (wet and dry) or non obstructive urinary retention who are therapy resistant to pelvic floor physiotherapy and medical management and wish to undergo a tined lead procedure.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
EMG pelvic floor | 1 day
  Latency and amplitude measured by probe

SECONDARY OUTCOMES:
Prevalence of adverse events | 2 years
  Prevalence of adverse events, which are defined as: pain, decrease in efficacy and number of reprogramming sessions.
Voiding diary | 1 year
  Determine the success rate of tined lead test period based upon changes in 3 days.
Validated questionnaires (KHQ and PeLFis) | 1 year
  Determine the success rate of tined lead test period based upon changes in validated questionnaires (KHQ and PeLFis).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan De Wachter, MD PhD FEBU, Study Director — University Hospital, Antwerp; Donald Vaganée, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No